CLINICAL TRIAL: NCT06280092
Title: A Pilot Study to Evaluate the Feasibility and Safety of Allogenic Adipose-derived Mesenchymal Stem Cells(AMSCs) for Epilepsy During Deep Brain Stimulation(DBS) Surgery
Brief Title: Allogenic Adipose-derived Mesenchymal Stem Cells(AMSCs) for Epilepsy During Deep Brain Stimulation(DBS) Surgery
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sanjeet S. Grewal (Other)
Responsible Party: Sponsor-Investigator, Sanjeet S. Grewal, Sponsor-Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-009133
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: A single dose of 5x10^6 AMSCs will be resuspended in 1ml of LRS and infused via intraparenchymal at the time of DBS surgery
Masking Description: This is an unmasked study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AMSCs (Experimental): A single dose of 5x10^6 AMSCs will be resuspended in 1ml of LRS and infused via intraparenchymal at the time of DBS surgery
  Interventions: Drug: AMSCs

INTERVENTIONS:
Drug: AMSCs — A single dose of 5x10^6 AMSCs will be resuspended in 1ml of LRS and infused via intraparenchymal at the time of DBS surgery

SUMMARY:
This study is a non-randomized, open label, phase 1 clinical trial to evaluate the fesibility and safety of intrathalamic delivery of MSCs during standard of care DBS surgery for epilepsy.

Subjects will be screened at our outpatient clinic and interested qualified subjects will be consented and offered participation in this trial. Once consent has been obtained, patients will undergo a standard preoperative evaluation which includes baseline laboratory values and a high-definition MRI. Patients will then undergo a stereotactic procedure for bilateral thalamic implantation of DBS leads through the ClearPoint® system. After the thalamic target for DBS is identified, cells will be infused directly into the anterior nucleus of the thalamus previous to lead implantation.

Patients will be followed in the outpatient setting for up to a year after therapy application.

Surgical, clinical, and radiographic data will be obtained during these visits

DETAILED DESCRIPTION:
To investigate the feasibility and safety of local delivery of AMSCs for epilepsy by measuring the incidence of AEs related to the study agent.

To investigate the effects of local delivery of AMSCs for epilepsy as measured by radiographic data on MRI.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥ 18 years of age.
* Participants with Drug Resistance Epilepsy as defined by the ILAE5.
* Participants undergoing bilateral implantation of DBS leads into the anterior nucleus of the thalamus.
* Adequate organ function as assessed by the following laboratory values within 3 weeks prior to admission to the study:
* Serum creatinine and urea < 2 times the upper limit of normal;
* ALT, AST and alkaline phosphatase < 3 times the upper limit of normal, and bilirubin < 2.5 mg/dL;
* Prothrombin time ≤ 1.5 times upper limit of normal;
* INR and PTT ≤ 1.5 times the upper limit of normal;
* Hemoglobin ≥ 9 g/dL;
* Platelets ≥ 100 x 10^9/L;
* Absolute Neutrophil Count (ANC) ≥ 1.5 x 10^9/L.
* Patient or legal guardian is able to fully understand and provide written and verbal consent for the protocol.
* Patient is a candidate for ANT DBS based on the following criteria established by the American Society for Stereotactic and Functional Neurosurgeons:
* Confirmed diagnosis of epilepsy by an epileptologist with focal-onset seizures, with or without generalization;
* Failure to adequately control seizures after two (or more) appropriate and adequately-dosed anti-seizure medications;
* Either partial-onset seizures with a localized onset in a region not amenable to resection or following failed resective surgery or focal-onset seizures with distributed or unclear onset zone.

Exclusion Criteria:

* Patients who have undergone a prior intracranial procedure for epilepsy.
* Patients with an intracranial tumor.
* Confirmed pregnancy.
* History of cancer not in remission for at least 5 years.
* History of diabetes, chronic renal failure, or other significant underlying medical or ----immunosuppressive conditions.
* History of drug or alcohol abuse.
* Subjects allergic to any component of the investigational product.
* Subjects > 75 years of age.
* Cognitively impaired adults.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs related to the study agent | 12 months
  To investigate the feasibility and safety of local delivery of AMSCs for epilepsy by measuring the incidence of AEs related to the study agent.
Radiographic effects related to the study agent | 12 months
  To investigate the effects of local delivery of AMSCs for epilepsy as measured by radiographic data on MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeet Grewal, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No